CLINICAL TRIAL: NCT07012668
Title: Outcomes and Risk Factors of Different Treatment Strategies for Neuro-co-cardiological Diseases and Post-cardiac Surgery Cerebrovascular Diseases
Status: Recruiting | Type: Observational
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Xiaochuan Huo, Prof, Beijing Anzhen Hospital
Other Study IDs: ANGEL-NEUROCARD
Record Dates: First submitted 2025-06-01; First posted 2025-06-10 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Neuro-co-cardiological Diseases; Post-cardiac Surgery Cerebrovascular Diseases; Vascular Lesion
Keywords: Neuro-co-cardiological diseases; Post-cardiac surgery Cerebrovascular diseases; Simultaneous treatment; Staged treatment; Conservative treatment
MeSH Terms: interventions — Methods; Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Neuro-co-cardiological diseases: Simultaneous treatment: Simultaneous interventional therapy/Simultaneous surgical treatment/ Simultaneous hybrid surgical treatment
  Interventions: Procedure: Interventional or surgical treatment
- Neuro-co-cardiological diseases: Staged treatment: Staged interventional therapy/Staged surgical treatment/Staged hybrid surgical treatment
  Interventions: Procedure: Interventional or surgical treatment
- Neuro-co-cardiological diseases: Conservative treatment: Surgery/intervention for one disease and conservative treatment for another disease or Simultaneously conservative treatment
- Post-cardiac surgery Cerebrovascular disease: Surgery/Interventional Treatment: Post-cardiac surgery Cerebrovascular disease: Surgery/Interventional Treatment
  Interventions: Procedure: Interventional or surgical treatment
- Post-cardiac surgery Cerebrovascular disease: Conservative treatment: Post-cardiac surgery Cerebrovascular disease: Conservative treatment

INTERVENTIONS:
Procedure: Interventional or surgical treatment — Simultaneous interventional or surgical treatment/staged interventional or surgical treatment
  Groups: Neuro-co-cardiological diseases: Simultaneous treatment; Neuro-co-cardiological diseases: Staged treatment
Procedure: Interventional or surgical treatment — Interventional or surgical treatment
  Groups: Post-cardiac surgery Cerebrovascular disease: Surgery/Interventional Treatment

SUMMARY:
The objective of this observational cohort study is to evaluate the clinical outcomes of various treatment strategies for cerebrovascular and cardiovascular diseases. Furthermore, it aims to investigate the factors that influence adverse outcomes from these treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years;
2. Patients with neuro-co-cardiological diseases or post-cardiac surgery cerebrovascular diseases.

Exclusion Criteria:

1. The expected survival is less than 1 years;
2. Simultaneously merge other serious diseases;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with neuro-co-cardiological diseases or post-cardiac surgery cerebrovascular diseases
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-09-19 (Actual); Primary Completion 2027-09-19 (Estimated); Study Completion 2027-09-19 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Scale Score | 90±7 days
  Modified Rankin Scale（0-6）, A lower MRS score indicates better functional status for the patient.

SECONDARY OUTCOMES:
Modified Rankin Scale Score | 7±1 days or the day discharged
  Modified Rankin Scale（0-6）, A lower MRS score indicates better functional status for the patient.
Modified Rankin Scale Score | 365±30 days
  Modified Rankin Scale（0-6）, A lower MRS score indicates better functional status for the patient.
Perioperative complication rate | 30±7 days
Rate of cardiovascular and cerebrovascular events | 90±7 days
Rate of cardiovascular and cerebrovascular events | 365±30 days
Short-term complications | 90±7 days
Long-term complications | 365±30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No